CLINICAL TRIAL: NCT05401565
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled, Two-Arm, Parallel-Group, Multicenter Study To Evaluate The Efficacy And Safety Of Balovaptan In Adults With Post-Traumatic Stress Disorder
Brief Title: Study To Evaluate The Efficacy And Safety Of Balovaptan In Adults With Post-Traumatic Stress Disorder (PTSD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BN43546
Record Dates: First submitted 2022-05-29; First posted 2022-06-02 (Actual); Results first posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-03

CONDITIONS: Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — balovaptan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Balovaptan (Experimental)
  Interventions: Drug: Balovaptan
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Balovaptan — Intervention of oral administration of 10mg balovaptan QD for 12 weeks followed by two weeks of follow-up period
  Arms: Balovaptan
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of 10 mg of oral administration balovaptan once a day (QD) compared with matching placebo in adults with PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have a current diagnosis of PTSD as per DSM-5 criteria, with a score of >/=33 on the PCL-5 at screening
* The index trauma event must have occurred in adulthood, i.e., when the participant was >/=18 years old
* The index trauma event must have occurred at least 6 months prior to screening and no more than 10 years prior to screening
* At baseline, either taking a stable dose of a single antidepressant (SSRI or SNRI) for management of PTSD and have been on that medication for >/=6 weeks at that stable dosage and demonstrating residual symptoms of PTSD or prior demonstrated lack of tolerability or lack of efficacy and not taking an antidepressant medication at baseline for >/=6 weeks
* Treatment with permitted medications and/or non-pharmacological interventions at a stable dose for 6 weeks prior to screening
* For women of childbearing potential: agreement to remain abstinent or use contraception

Exclusion Criteria:

* Participants who are experiencing ongoing exposure to traumatic events within 3 months of screening
* Participants who are pregnant or breastfeeding, or intending to become pregnant during the study or within 14 days after the final dose of study drug
* Clinically significant psychiatric and/or neurological conditions, which may interfere with the assessment of safety or efficacy endpoints
* Substance use disorders during last 12 months
* Significant risk for suicidal behaviour
* Epilepsy or seizure disorder considered not well controlled within the past 6 months or changes in anticonvulsive therapy within the last 6 months
* Clinical diagnosis of peripheral neuropathy
* Within the last 2 years, unstable or clinically significant cardiovascular disorders
* Positive serology results for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) 1 or 2
* Moderate or severe hepatic or renal impairment
* History of coagulopathies, bleeding disorders, blood dyscrasias, hematological malignancies, myelosuppression (including iatrogenic)
* Medical history of malignancy, if not considered cured
* Participants who have received treatment with investigational therapy within 8 weeks prior to randomization
* Known hypersensitivity to balovaptan, its components, or any of the excipients used in the formulation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2023-10-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Alea Research, Phoenix, Arizona
  - CITrials, Inc., Bellflower, California
  - ASCLEPES Research Centers, Panorama City, California
  - Clinical Innovations, Inc, Santa Ana, California
  - Sarkis Clinical Trials, Gainesville, Florida
  - Galiz Research, LLC, Hialeah, Florida
  - Florida International Research Center, Miami, Florida
  - American Medical Research, Inc, Oak Brook, Illinois
  - Boston Clinical Trials & Medical Research, Roslindale, Massachusetts
  - Michigan Clinical Research Institute PC - Clinedge - PPDS, Ann Arbor, Michigan
  - Va Medical Center, Minneapolis, Minnesota
  - Alivation Research, LLC, Lincoln, Nebraska
  - Bioscience Research, LLC, New York, New York
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Donald J. Garcia Jr., MD, PA, Austin, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: More participants (29) were enrolled than initially planned (16)
Period: Overall Study
Arm/Group | Placebo | Balovaptan
Started | 16 | 13
Completed | 13 | 13
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Balovaptan | Total
Number analyzed (Participants) | 16 | 13 | 29
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.6 (8.2) | 38.2 (13.8) | 37.3 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 13 | 10 | 23
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Clinician-Administered PTSD Total Symptom Severity Score
Description: The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) measures the severity of PTSD where smaller scores indicate less severe PTSD and higher scores suggest more severe PTSD. Possible scores for this 30 item version range from 0 to 120. Measured 3 times over 12 weeks.
Time Frame: From Baseline up to Week 12
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Placebo | Balovaptan
Number analyzed (Participants) | 16 | 13
Score on a Scale
  Baseline | 35.5 (9.3) | 33.8 (7.8)
  Week 6: number analyzed (Participants) | 13 | 13
  Week 6 | -6.8 (11.2) | -10.3 (9.2)
  Week 12: number analyzed (Participants) | 12 | 13
  Week 12 | -15.6 (10.6) | -17.2 (10.7)

2. Secondary Outcome: Symptom Severity as Measured by Clinician-Global Impression of Severity (CGI-S) Scale Score
Description: The CGI-S reflects the rater's impression of the subject's current PTSD severity on a 6-point scale ranging from no symptoms (1) to very severe symptoms (6).
Time Frame: From Baseline up to Week 12
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Balovaptan
Number analyzed (Participants) | 16 | 13
Participants
  Baseline Very mild: number analyzed (Participants) | 15 | 13
  Baseline Very mild | 0 | 0
  Baseline Mild: number analyzed (Participants) | 15 | 13
  Baseline Mild | 1 | 0
  Baseline Moderate: number analyzed (Participants) | 15 | 13
  Baseline Moderate | 3 | 8
  Baseline Severe: number analyzed (Participants) | 15 | 13
  Baseline Severe | 11 | 5
  Baseline Very severe: number analyzed (Participants) | 15 | 13
  Baseline Very severe | 0 | 0
  Week 6 Very mild: number analyzed (Participants) | 12 | 13
  Week 6 Very mild | 0 | 0
  Week 6 Mild: number analyzed (Participants) | 12 | 13
  Week 6 Mild | 0 | 4
  Week 6 Moderate: number analyzed (Participants) | 12 | 13
  Week 6 Moderate | 4 | 8
  Week 6 Severe: number analyzed (Participants) | 12 | 13
  Week 6 Severe | 8 | 1
  Week 6 Very severe: number analyzed (Participants) | 12 | 13
  Week 6 Very severe | 0 | 0
  Week 12 No Symptoms: number analyzed (Participants) | 13 | 13
  Week 12 No Symptoms | 2 | 0
  Week 12 Very mild: number analyzed (Participants) | 13 | 13
  Week 12 Very mild | 0 | 1
  Week 12 Mild: number analyzed (Participants) | 13 | 13
  Week 12 Mild | 3 | 6
  Week 12 Moderate: number analyzed (Participants) | 13 | 13
  Week 12 Moderate | 5 | 5
  Week 12 Severe: number analyzed (Participants) | 13 | 13
  Week 12 Severe | 3 | 1
  Week 12 Very severe: number analyzed (Participants) | 13 | 13
  Week 12 Very severe | 0 | 0

3. Secondary Outcome: Change From Baseline at Week 12 in the Patient Health Questionnaire-9 (PHQ-9) Total Score
Description: PHQ-9 is a 9-item PRO used to assess severity of depression. Responses are rated based on frequency of symptoms on a 4-point Likert scale, ranging from 0 (not at all) to 3 (nearly every day). A total PHQ-9 total score ranging from 0 to 27 can be calculated by summing the nine items, of which a higher score corresponds to more severe depression.
Time Frame: From Baseline up to Week 12
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Placebo | Balovaptan
Number analyzed (Participants) | 16 | 13
Score on a Scale
  Baseline: number analyzed (Participants) | 15 | 13
  Baseline | 15.2 (4.8) | 12.2 (5.1)
  Week 6: number analyzed (Participants) | 14 | 13
  Week 6 | -2.7 (5.6) | -2.5 (5.8)
  Week 12: number analyzed (Participants) | 13 | 13
  Week 12 | -6.0 (5.1) | -3.5 (5.2)

4. Secondary Outcome: Percentage of Participants With Adverse Events
Time Frame: From Baseline up to Week 12
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Balovaptan
Number analyzed (Participants) | 16 | 13
Participants | 7 | 9

ADVERSE EVENTS:
Time Frame: Up To 12 Weeks
Groups:
- BALOVAPTAN 10 MG: ntervention of oral administration of 10mg balovaptan QD for 12 weeks followed by two weeks of follow-up period
Arm/Group | PLACEBO | BALOVAPTAN 10 MG
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/13
Other Adverse Events (participants affected / at risk) | 7/16 | 9/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLACEBO (N=16) | BALOVAPTAN 10 MG (N=13)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0)
Muscle contractions involuntary (Nervous system disorders) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0)
Libido decreased (Psychiatric disorders) | 0 (0) | 0 (0)
Mood swings (Psychiatric disorders) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLACEBO (N=16) | BALOVAPTAN 10 MG (N=13)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 1 (1)
Muscle contractions involuntary (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Libido decreased (Psychiatric disorders) | 1 (1) | 0 (0)
Mood swings (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-09): https://cdn.clinicaltrials.gov/large-docs/65/NCT05401565/Prot_SAP_000.pdf